CLINICAL TRIAL: NCT04402723
Title: A Dose-escalated Phase Ⅰ Trial to Assess the Tolerance and Pharmacokinetics of Combination of Donafenib and Cytarabine/Daunorubicin in Relapsed AML Patient
Brief Title: Combination of Donafenib and Cytarabine/Daunorubicin in Relapsed AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate policy adjustments
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZGDAML1
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — donafenib; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donafenib, 0.2g (Experimental): Donafenib,0.2g,bid,Combination with Cytarabine and Daunorubicin.
  Interventions: Drug: Donafenib
- Donafenib,0.3g (Experimental): Donafenib,0.3g,bid,Combination with Cytarabine and Daunorubicin
  Interventions: Drug: Donafenib

INTERVENTIONS:
Drug: Donafenib — In first 28-days-cycle, eligible subjects will be given Donafenib 0.2/0.3g, bid, for first 14 days, combination with Daunorubicin 60mg/m2/d, for first 3 days, and Cytarabine 100mg/m2/d, for first 7 days. If CR or CRi is observed, subjects will be given Donafenib 0.2/0.3g, bid, for first 14 days, combination Cytarabine 2g/m2/q12h, for first 3 days, in next 28-day-cycle.
  Other Names: Cytarabine and Daunorubicin

SUMMARY:
This phase Ⅰ study of Donafenib, an oral multikinase inhibitor that targets Raf kinase and receptor tyrosine kinases, is to assess safety and pharmacokinetics in patients with Relapsed AML.

DETAILED DESCRIPTION:
Donafenib is a multikinase inhibitor which is acting on various cellular pathways involved in the genesis of acute myeloid leukemia (AML). Donafenib is therefore a promising candidate for improvement of chemotherapy results in AML. This clinical trial evaluates the safety and pharmacokinetics of Donafenib combination with Cytarabine/Daunorubicin for AML in patients between 18 and 55 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed AML (except APL) according to the FAB and WHO classification, including AML evolving from MDS or other hematologic diseases and AML after previous cytotoxic therapy or radiation (secondary AML) .
* Patients with diagnosed Relapsed AML according to Chinese Guidelines for the Diagnosis and Treatment of Acute Myeloid Leukemia.
* relapse after 6 months of an morphological remission.
* Age ≥ 18 and ≤ 55 years.
* BMI ≥ 18 and ≤27.
* Informed consent, personally signed and dated to participate in the study.
* ECOG performance status of 0-1.
* Life expectancy of at least 12 weeks.
* Total serum bilirubin ≤1.5×ULN.
* Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5×ULN.
* Serum creatinine ≤1.5×ULN.
* glomerular filtration rate ≥60 mL/min, as calculated with the Cockcroft-Gault formula.
* alkaline phosphatase ≤1.5×ULN.
* urine protein ≤1+, or Urine protein was quantified for 24h ≤0.5g.
* INR/PTT <1.5×ULN.

Exclusion Criteria:

* Patients who are not eligible for standard chemotherapy as per discretion of the treating physician.
* Patients who have been treated with bone marrow transplantation.
* Central nervous system manifestation of AML.
* Cardiac disease: heart failure NYHA III or IV; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Patients who have thrombosis events within 6 months prior to study entry is permitted.
* Pregnancy or breastfeed.
* Chronic pulmonary disease with relevant hypoxia.
* Patients undergoing dialysis.
* Known HIV and/or hepatitis C infection.
* Evidence or history of severe non-leukemia associated bleeding diathesis or coagulopathy.
* Evidence or recent history of CNS disease, including primary or metastatic brain tumors, seizure disorders.
* Blood pressure (BP) higher than systolic 140 mmHg and/or diastolic 90 mmHg after best treatment.
* Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance of the protocol.
* Patients with major surgery, open biopsy or significant traumatic injury within 4 weeks prior to study entry is permitted.
* Serious, non-healing wound, ulcer or bone fracture.
* Infection need antibiotic treatment.
* Cumulative therapeutic dose of Daunorubicin more than 300mg/m2.
* Concurrent malignancies other than AML.
* History of organ allograft.
* Allergy to study medication or excipients in study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Safety(including the type, severity and frequency of AE) | through study completion, an average of 2 months
  Safety of combination of donafenib with Cytarabine/Daunorubicin in relapsed AML patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Doctor, Principal Investigator — Institute of Hematology and Blood Disease Hospital
Locations (1):
- Institute of Hematology and Blood Disease Hospital, Tianjin, Tianjin Municipality, China